CLINICAL TRIAL: NCT05485909
Title: A Single-arm, Single-center Phase II Clinical Study of Regorafenib and Toripalimab Combined With Radiofrequency Ablation (RFA) in Patients With Colorectal Cancer Liver Metastases
Brief Title: Phase II Study of Regorafenib and Toripalimab Combined With RFA in Patients With CRCLM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhiqing Wang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-319-003
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer Liver Metastases
MeSH Terms: interventions — Radiofrequency Ablation; regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib and Toripalimab Combined with RFA (Experimental)
  Interventions: Other: Radiofrequency ablation; Drug: Regorafenib and Toripalimab Combination

INTERVENTIONS:
Other: Radiofrequency ablation — For multiple intrahepatic lesions, select 1 to 2 lesions for radiofrequency ablation
Drug: Regorafenib and Toripalimab Combination — Toripalimab 200 mg, iv drip, d1, d15, q4w, Regorafenib 80mg, po, d1-d21, Q4w.

SUMMARY:
The incidence of colorectal cancer liver metastasis is high and the prognosis is poor. Improving the treatment effect of colorectal cancer liver metastasis is the key to improving the prognosis of colorectal cancer patients. Rigofenib is one of the standard third-line treatments for advanced colorectal cancer, but has limited efficacy. Immune checkpoint inhibitors (PD-L1 monoclonal antibody, PD-1 monoclonal antibody) have achieved good results in the treatment of various malignant tumors. In a mouse transplant tumor model of colorectal cancer, regorafenib combined with PD-1 monoclonal antibody treatment significantly improved the antitumor activity, but the efficacy rate in clinical studies was not very high, especially for liver metastases. Radiofrequency ablation (RFA) is one of the common methods for the treatment of liver metastases. RFA may improve the immune microenvironment and the efficacy of immunotherapy,and the purpose of this trial is to explore the efficacy and safety of rigofenib and terepliumab combined with RFA in patients with refractory colorectal cancer liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years;
2. Histologically or cytologically confirmed colon or rectal adenocarcinoma, with unresectable relapsed or metastatic disease;
3. Microsatellite stability (MSS) or microsatellite instability-low (MSI-L), or proficient expression of DNA mismatch repair gene (pMMR);
4. Patients who have failed, or can not tolerate after previous systemic treatment for relapsed or metastatic colorectal cancer, with no more than 3 months for disease progression after the last systemic treatment. The systemic treatment must contain fluorouracil, oxaliplatin and irinotecan, with or without targeted therapy (bevacizumab, cetuximab, and so on);
5. According to the RECIST 1.1 standard, in addition to the lesion to be ablated and the measurable lesion outside the liver, there is at least one measurable lesion in the liver. Measurable lesions were defined as non-lymph node lesions with the longest single diameter ≥ 10 mm, or lymph node lesions with a short diameter ≥ 15 mm;
6. ECOG score 0-1;
7. Expected survival ≥3 months;
8. Good organ function (without blood transfusion, use of hematopoietic stimulating factors, or transfusion of albumin or blood products within 14 days prior to examination):

1）Platelet (PLT) count ≥100,000 /mm3; 2) Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6) Total bilirubin (TBIL) level ≤1.5×ULN; 7) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 8) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 9) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min; 10) Thyroid stimulating hormone (TSH) ≤ULN; 11) Normal serum free thyroid hormone (T4); 12) Normal serum free triiodothyronine (T3); 13) Serum amylase ≤1.5×ULN; 15) Lipase ≤1.5×ULN.

9. Females of child bearing age must have a negative pregnancy test, and have to take contraception measures and avoid breast feeding during the study and for 3 months after the last dose; male subjects must agree to taken contraception measures during the study and for 3 months after the last dose.

10. Able to understand and willing to sign written informed consent form.

Exclusion Criteria:

1. Diagnosis of any other malignancy at different primary site or of different histological type from colorectal cancer within 5 years prior to initiation of study treatment, except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of cervix;
2. Microsatellite instability-high (MSI-H) or deficient expression of DNA mismatch repair gene (dMMR);
3. Previous treatment with regorafenib, PD-1/PD-L1/PD-L2 antibody or any other antibody that acts on T cell costimulatory or checkpoint pathways;
4. Known allergy to study drug or excipients, or allergy to similar drugs;
5. Have received other anti-tumor treatment within 4 weeks prior to initiation of study treatment, or no more than 5 half lives from the last dose;
6. Have participated in other clinical study and received drug within 4 weeks prior to initiation of study treatment;
7. Have undergone major surgery or open biopsy, or have massive trauma within 4 weeks prior to initiation of study treatment;
8. Have received immunosuppressants (excluding inhaled corticosteroids or ≤10 mg/day prednisone or other systemic steroids at equivalent pharmaphysiological dose) within 2 weeks prior to initiation of study treatment;
9. Have vaccination with attenuated live vaccines within 4 weeks prior to initiation of the study treatment or plan to vaccinate during the study;
10. CYP3A4 inducers or inhibitors should not be stopped within 1 week prior to initiation of study treatment and during the study;
11. Known metastasis to central nervous system;
12. Present or history of any autoimmune disease;
13. Human immunodeficiency virus (HIV) infection (HIV antibody positive), or active hepatitis C virus (HCV) infection (HCV antibody positive), or active hepatitis B virus (HBV) infection (HBsAg or HBcAb positive, and HBV-DNA ≥2000 IU/ml (copies/ml)), or other severe infection requiring systemic antibiotic treatment, or unexplained body temperature >38.5℃ during screening period/before study treatment;
14. Presence of pleural effusion, peritoneal effusion, or pericardial effusion;
15. Development of the following diseases within 6 months prior to initiation of study treatment: myocardial infarction, severe/unstable angina, congestive heart failure above NYHA grade 2, poorly controlled arrhythmia;
16. Poorly controlled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
17. With bleeding tendency, or evident hemoptysis or other hemorrhagic events (e.g. gastrointestinal hemorrhage, hemorrhagic gastric ulcer) within 2 months prior to initiation of study treatment, or presence of hereditary or acquired bleeding or thrombotic tendency (e.g. hemophilia, coagulopathy, thrombocytopenia, etc.), or current/long-term thrombolytic or anticoagulant therapy (except aspirin ≤100 mg/day);
18. Development of arterial/venous thrombotic events, e.g. cerebrovascular accident (transient ischemic attack, cerebral hemorrhage, cerebral infarction etc.), deep venous thrombosis, vasculitis, etc. within 6 months prior to initiation of study treatment;
19. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
20. Seizure requiring drug (e.g. steroids or antiepileptic drugs) treatment;
21. Presence of malabsorption disorder;
22. Unable to swallow study drug;
23. Presence of toxicities (except alopecia) of grade 2 and above (CTCAE V5.0) due to previous anti-tumor treatment or surgical procedure;
24. History of drug abuse, illegal drug use or alcohol dependence;
25. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The ratio of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Time from first dose to first documented disease progression or death from any cause (whichever occurs first)
Overall survival (OS) | 2 years
  Overall survival (OS) was defined as the time (days) from randomization to death due to any cause.
Disease control rate (DCR) | 2 years
  Defined as the proportion of patients whose tumors shrink or remain stable for a certain period of time, including CR, PR and SD
Duration of response (DOR) | 2 years.
  defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death
Time to disease progression (TTP) | 2 years
  Time from first dose to first documented disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiqiang Wang, Guangzhou, Other (Non U.s.), China